CLINICAL TRIAL: NCT05987657
Title: Comparison of Two Methods to Assess Progesterone Concentration in Patient During IVF Protocol on Triggering Day: Salivary Versus Blood Test
Brief Title: Assessment of Two Methods for Progesterone Dosage During IVF
Acronym: SALIPROG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL23_0644
Record Dates: First submitted 2023-07-28; First posted 2023-08-14 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Infertility
Keywords: Progesterone concentration; salivary test; In vitro fertilization; infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Salivary and blood progesterone dosage (Other): IVF patients with fresh embryo transfer having a dosage of progesterone, salivary and blood, on triggering day
  Interventions: Diagnostic Test: Salivary and blood progesterone dosage

INTERVENTIONS:
Diagnostic Test: Salivary and blood progesterone dosage — Salivary dosage: patient will chew a dry swab for 2 minutes; when the swab is soaked it is put back in its small case and sent to the laboratory for analysis.
  In parallel, the same patients will have a blood sample of 4 ml to dose blood progesterone on an EDTA tube. It will be also sent to the laboratory for analysis.
  Both analyses will be done only once on triggering day meaning 36 hours before oocyte retrieval.

SUMMARY:
Nowadays, 1/7 couple consult because of infertility and some of them will need in vitro fertilization +/- intracytoplasmic sperm injection (IVF+/- ICSI). The IVF process includes a 14 days stimulation with FSH +/- LH in an agonist or antagonist protocol. The monitoring consists of regular ultrasound scan and blood sample. During the stimulation protocol many test have been proposed to predict the success of IVF. However, progesterone dosage on triggering day seems to be the only relevant exam. Indeed, when the progesterone blood concentration is low, the pregnancy rate is decreased. The only way to obtain progesterone concentration is a blood sample. The IVF journey is known to be stressful with many injections. Therefore, the salivary dosage appear to be more patient friendly. This kind of dosage has already been studied yet never use in routine because of a lack of repeatability. The laboratory of Lyon has developed a new technique to overcome this issue by using a liquid chromatography-mass spectrometry.

The aim of this work is as a first step to assess the repeatability, reliability and precision of salivary dosage on triggering day for IVF patient compared to blood concentration of progesterone.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients between 18 and under 43 years old
* in the course of IVF more or less ICSI of the PMA service of the HFME with transfer of fresh embryo
* Signature of an express consent
* Understanding the French language, both oral and written.
* Affiliated to a social security scheme

Exclusion Criteria:

* Persons deprived of their liberty by a judicial or administrative decision
* Persons subject to psychiatric care
* Persons admitted to a health or social establishment for purposes other than research
* Participants in another study that could impact the results of the present study, in particular those related to the level of progesterone.
* Adults subject to a legal protection measure (guardianship, curatorship)

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-11-09 (Actual); Study Completion 2024-11-09 (Actual)

PRIMARY OUTCOMES:
Reliability of salivary dosage of progesterone compared to blood sample. | At the inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Femme Mère Enfant, Bron, Rhône, France

IPD SHARING:
Plan to Share IPD: No